CLINICAL TRIAL: NCT04366804
Title: International Validation of Two Non-motor Scales in Parkinson's Disease: the Neuropsychiatric Fluctuations Scale (NFS) and the Shame in Parkinson's Disease (SPARK) Scale
Brief Title: International Validation of Two Non-motor Scales in PD (NFS and SPARK)
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-00303
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease; Non-motor Symptoms
Keywords: Parkinson's Disease; Non-motor symptoms; Scales for non-motor symptoms; Validation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with neuropsychiatric fluctuations: PD patients with neuropsychiatric fluctuations (≥ 2 positive answers in QUICK test)
- Patients without neuropsychiatric fluctuations: PD patients without neuropsychiatric fluctuations (≤ 1 positive answer in QUICK test)

SUMMARY:
The goal of this project is to develop the international validation of two new rating scales, the Neuropsychiatric Fluctuations Scale (NFS) and the Shame in PARKinson's disease (SPARK) Scale, in order to improve the understanding of the extent and severity of non-motor symptoms in Parkinson's disease (PD).

DETAILED DESCRIPTION:
This project is a prospective international multicentre study to validate two new rating scales in different languages: the Neuropsychiatric Fluctuations Scale (NFS) and the Shame in PARKinson's disease (SPARK) Scale.

The project population consists a minimum of 300 PD patients with and without fluctuations in the participant countries: Spain, Germany, France, Switzerland, Romania and Greece.

The NFS is specifically designed to detect neuropsychiatric fluctuations between off- and on-medication condition in PD. It is composed of 20 items, 10 items measuring the on-neuropsychological symptoms and 10 items for the off-neuropsychological manifestations. The validation of this scale, based on the most frequently experienced symptoms by the patients, would allow a crucial breakthrough in the improvement of management of PD patients.

Shame and embarrassment are poorly recognized by physicians in PD. PD-related shame and embarrassment may emerge from motor and non-motor symptoms, from self-perception of inadequacy due to loss of autonomy and need for help, or from perceived deterioration of body image. The current available scales are not specific for PD. Based on reports of persons affected with PD and a literature review about shame and stigmatization in PD a 25-items self-questionnaire for shame and embarrassment in PD was created. The scale includes 6 different subscales (1. Shame arising from PD symptoms; 2. Shame arising from the increasing physical dependence and need for help induced by PD; 3. Shame arising from the patient's assumption of breaking certain social rules; 4. Shame arising from the deteriorated body image; 5. Consequence of related shame and embarrassment on patients' health-related quality of life; 6. Stigmatization). The validation of this scale will give a tool for physicians and researchers to better understand the impact of PD on patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. PD, according to the MDS criteria;
3. Age of participants > 30 and < 75 years;
4. Being fluent in the language in which the scales are applied.

Exclusion Criteria:

1. Presence of PD dementia (defined as MoCA score < 24).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project population consists of PD patients with and without neuropsychiatric fluctuations attending routine visits to movement disorders clinics in the participant countries. Only patients capable of giving informed consent will be considered for participation in this project.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NFS score | 2 weeks (2 assessments in a time span of 2 weeks)
SPARK score | 2 weeks (2 assessments in a time span of 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, MD, PhD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (8):
- Centre hospitalier régional universitaire de Besançon, Besançon, France
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Transilvania University, Brasov, Romania
- Spain (2):
  - Hospital Universitario Burgos, Burgos
  - Ruber International Hospital, Madrid
- Insel Gruppe AG University Hospital Bern, Bern, Switzerland
- King's College London, London, United Kingdom